CLINICAL TRIAL: NCT02147236
Title: A Randomized Trial of a Structured Social Skills Development Progam for Children With Autism Spectrum Disorders
Brief Title: Social Skills in Children With Autism Spectrum Disorders
Acronym: SSD_ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Organization of Autism Research (Unknown); Renfield Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0402026356
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Pervasive Developmental Disorders
Keywords: autism; pervasive developmental disorders; social skills intervention
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Social Skills Training

SUMMARY:
To evaluate whether a structured social skills program, called Social Skills Development,is superior to a wait list control group on measures of interpersonal interaction. The Social Skills Development (SSD) is a 16-week, group intervention that uses activities and peer tutors to promote interpersonal skills in children 8 to 11 years of age with Autism Spectrum Disorders.Following a diagnostic and social skills assessment,children are randomly assigned to SSD or wait list for 16 weeks. Children who were randomized to the wait list are offered SSD at Week 16. Children randomized to SSD are followed for 9 months to assess the durability of gains during the first 16 weeks.

DETAILED DESCRIPTION:
This project is designed to evaluate the acceptability and initial efficacy of a structured group treatment intervention for enhancing social behavior in 40 children with autism spectrum disorders (ASDs). An important long-term goal of this project was to develop a model for delivery of social skills training that could be tested in a larger trial and ultimately exported to schools and community settings. To accomplish these aims, we designed a randomized clinical trial to evaluate a structured social skills program for school age children with pervasive developmental disorders (PDDs)compared to a Wait List control group. Specific aims included gathering preliminary evidence on the efficacy of the intervention on various parent measures of behavior, as well as an assessment of overall social functioning by an independent rater who would be blind to treatment assignment. The Social Skills Development program uses semi-structured activities and peer tutors to promote interpersanal skills. To evaluate acceptability of the program, we planned to track attendance, attrition and parent satisfaction in the trial. Finally, to evaluate the durability of gains achieved during the Social Skills Development program, we re-assessed the subjects initially randomized to the active treatment group at 9 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 11 years
* Full Scale IQ score > 70
* PDD diagnosis (autism, Asperger's, PDD-Not Otherwise Specified)

Exclusion Criteria:

* concurrent, untreated psychiatric disorder(such as anxiety, depression or conduct disorder)

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2003-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression for Improvement | 16 weeks

SECONDARY OUTCOMES:
Social Competence Inventory | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D Scahill, MSN,PhD, Principal Investigator — Yale University Child Study Center
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States